CLINICAL TRIAL: NCT04508166
Title: Pharmacological Prevention of Post-traumatic Intrusions in Healthy Volunteers - Towards a Post-exposition Prophylaxis for Post-traumatic Stress Disorder
Brief Title: Towards a Post-exposition Pharmacological Prophylaxis for Post-traumatic Stress Disorder
Acronym: TRAUMA-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: TRAUMA-PROPHYLAXIS
Record Dates: First submitted 2020-07-31; First posted 2020-08-11 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Intrusive Thought; Psychological Trauma; Inflammatory Response; Physiological Stress
MeSH Terms: conditions — Psychological Trauma | interventions — Dexmedetomidine; Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine (Experimental): Sublingual dose of dexmedetomidine
  Interventions: Drug: Dexmedetomidine; Drug: Placebo; Behavioral: Experimental Model Trauma Film
- Gamma-hydroxybutyrate (Active Comparator): Oral dose of gamma-hydroxybutyrate
  Interventions: Drug: Gamma-Hydroxybutyrate; Drug: Placebo; Behavioral: Experimental Model Trauma Film
- Placebo (Placebo Comparator): Oral (saline) and sublingual (orodispersible tablet) doses
  Interventions: Drug: Dexmedetomidine; Drug: Placebo; Behavioral: Experimental Model Trauma Film

INTERVENTIONS:
Drug: Dexmedetomidine — Volunteers receive a single dose of dexmedetomidine sublingually at scheduled bedrest in the sleep laboratory
  Other Names: Dexdor
  Arms: Dexmedetomidine; Placebo
Drug: Gamma-Hydroxybutyrate — Volunteers receive a single oral dose of gamma-hydroxybutyrate at scheduled bedrest in the sleep laboratory
  Other Names: Xyrem
  Arms: Gamma-hydroxybutyrate
Drug: Placebo — Volunteers receive an oral (saline) or sublingual (orodispersible tablet) at scheduled bedrest in the sleep laboratory
Behavioral: Experimental Model Trauma Film — Each volunteer views experimental model trauma film before scheduled bedrest in the sleep laboratory. This video is ca. 15 minutes in duration and is composed of short (a few seconds to a few minutes) individual and unrelated scenes of violent death and injury of varying description. Six versions of the film without re-occurring scenes will be presented in balanced order across drug order conditions.

SUMMARY:
In this study, we investigate the role that deep sleep plays in the prevention of posttraumatic stress disorder after someone has been exposed to a trauma by boosting deep sleep with two drug conditions compared to placebo condition. Each volunteer in the study goes through all three conditions. The quantity of intrusive memories of the trauma will be compared between the three conditions.

DETAILED DESCRIPTION:
The present study seeks to investigate the potential to pharmacologically modulate slow-wave sleep in the acute aftermath of an experimentally-induced trauma in the interest of developing a secondary prevention of posttraumatic stress disorder. The effects of a GABAergic compound will be compared with that of a noradrenergic compound. Memory, sleep and stress-related immune response factors will be quantified and compared across drug conditions.

ELIGIBILITY:
Inclusion Criteria:

* Speaks and understands German
* BMI 18.5 -< 25
* Non-smoker status
* Habitual 5 or fewer alcoholic beverages / week
* Habitual 3 or fewer caffeinated beverages / day
* Habitual average sleep duration 7-9 h / night
* Normal or corrected-to-normal vision
* Insomnia Severity Index score between 8-14

Exclusion Criteria:

* Travel across 3 or more time zones within 3 months of study start
* Habitual napping
* Extreme chronotype, determined by Morningness-Eveningness Questionnaire
* History of or presence of a trauma- or stressor-related disorder
* History of or presence of neurological disorder, psychiatric disorder or head injury
* History of or presence of a sleep disorder
* History of or presence of cardiovascular disorder
* Use of illicit drugs
* Atypical preference for excessively violent portrayals
* Faints at the site of blood or brutality
* Has participated in a study < 30 days or a study such as this (i.e., experimental trauma) at all.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
Frequency of intrusive memories | Three weeks
  The number of intrusive memories of the experimental model trauma film experienced. The number of intrusive memories will be recorded in a diary by participants.
Emotional valence of intrusive memories | Three weeks
  The emotional valence will be recorded in a diary after experiencing an intrusive memory in an integer scale. The integer scale will range from 1 to 10, where 1 indicates the lowest and 10 indicates the highest.
Personal significance of intrusive memories | Three weeks
  Personal significance of intrusive memories will be recorded in a diary after experiencing an intrusive memory in an integer scale. The integer scale will range from 1 to 10, where 1 indicates the lowest and 10 indicates the highest.
Oscillatory delta power in the sleep electroencephalogram (EEG) during non rapid eye movement (REM) sleep stages N2 and N3 | Four nights, each night a week apart, spanning one month
  Power in units microvolts squared will be quantified by fast Fourier transform in 4 second segment length in EEG sleep recordings in the delta frequency bin (0.5 - 4.5 Hz).Higher value of delta power indicates greater homeostatic sleep pressure, i.e., the feeling of need for sleep.
Oscillatory theta power in the sleep electroencephalogram (EEG) during non rapid eye movement sleep stages N2 and N3 | Four nights, each night a week apart, spanning one month
  Power in units microvolts squared will be quantified by fast Fourier transform in 4 second segment length in EEG sleep recordings in the theta frequency bin (6 - 9 Hz). Higher value of theta power indicates greater homeostatic sleep pressure, i.e., the feeling of need for sleep.
EEG measures of sleep quality: distribution of N2 and N3 sleep stages. | Four nights, each night a week apart, spanning one month
  Number of non-REM sleep stages N2 and N3. Greater number of stages N2 and N3 indicate greater homeostatic sleep pressure, i.e., the feeling of need for sleep.
EEG measures of sleep quality: number of arousals | Four nights, each night a week apart, spanning one month
  Number of arousals Arousals are defined by the American Academy of Sleep Medicine as an increase in EEG frequency at least 3 seconds in NREM sleep in alpha, theta or higher frequencies, excluding spindles; must be accompanied by a minimum of 1 second of muscle activity during REM sleep. The greater the number of arousals indicates the lower homeostatic sleep pressure is in healthy individuals. Normal number of arousals for a healthy adult is ca. 80 per 8 hour sleep episode.
EEG measures of sleep quality: sleep onset latency | Four nights, each night a week apart, spanning one month
  Sleep onset latency represents elapsed time from intention to initiate sleep until sleep is initiated (defined as the occurrence of any stage of sleep by the AASM). Longer latencies indicate lower homeostatic sleep pressure or some maladaptive, e.g., rumination, stress, or pathological state, e.g., insomnia, posttraumatic stress. Normal latencies for healthy adults is 10 - 20 minutes.
EEG measures of sleep quality: sleep duration | Four nights, each night a week apart, spanning one month
  Sleep duration represents the duration in time of a sleep episode excluding any intervening stages of waking. Typical sleep duration in the healthy adult population is ca. 8 hours. Extreme sleep durations (<5 or <6 hr or >10 hr) have been associated with cardiometabolic illness risk.
EEG measures of sleep quality: sleep efficiency | Four nights, each night a week apart, spanning one month
  Sleep efficiency represents how efficient a given sleep episode is and is defined as the duration of sleep (i.e., time spent in all NREM and REM sleep stages) divided b by the total time spent in bed and multiplied by 100. Normal sleep efficiency is 80% or greater. Efficiencies less than this value could raise questions of sleep satiety, maladaptive behavior (e.g., alcohol consumption, caffeine consumption, sleep at incongruent circadian phase) or pathological health conditions (e.g., restless legs, disordered breathing, insomnia).

SECONDARY OUTCOMES:
Physiological stress: circulating cortisol | Four nights, each morning a week apart, spanning one month
  Cortisol (nmol/l) is a marker of stress activation and will be quantified by salivary assay. Greater values indicate greater stress response. Salivary cortisol concentrations vary by sex; in males it ranges under normal conditions from 1-50 nmol/l.
Physiological stress: electrocardiogram (ECG) heart rate (HR) | Four nights, each night a week apart, spanning one month
  Average resting ECG HR during waking in healthy adult males is 75 bpm (range: 60 - 100 bpm). Higher HR from an individual's baseline HR during and after experimental model trauma will be indicative of increases in sympathetic activation of heart function.
Physiological stress: respirometry respiration rate | Four nights, each night a week apart, spanning one month
  Resting respiration rate of an adult male is 12 - 16 breaths per minute. Increases in the number of breaths per minute will indicate increase in sympathetic activation of the autonomic system.
Physiological stress: electrocardiogram (ECG) heart rate variability (HRV) | Four nights, each night a week apart, spanning one month
  Heart rate variability will be quantified by measuring inter-beat intervals of the ECG. The normal-to-normal interval will be taken, which is the interpolated interval between normal R peaks of the QRS wave complex of the ECG. HRV values indicate performance of the autonomic nervous system in a given context. Higher values of sympathetic activation will be expected during experimental model trauma film exposure.
Physiological stress: inflammatory immune factors (cytokines and kynurenines) | Four mornings, each morning a week apart, spanning one month
  Lower concentration values of immune factors will be expected in GHB or DMTN conditions compared to placebo conditions.
Subjective ratings of mood: Positive and Negative Affect Scale (PANAS) | Four nights, each night a week apart, spanning one month
  The PANAS scale assesses affect and is comprised of a positive affect subscales and a negative affect subscale. The range of scores of either are 10 - 50. Higher scores in the positive subscale indicate higher (i.e., "better") mood; lower scores in the negative affect subscale indicate lower (i.e., "worse") mood. Mean (i.e., scores for normal healthy adults) respective scores for the positive and negative subscales are 33.3 (standard deviation [SD] = 7.2) and 17.4 (SD = 6.2).
Subjective ratings of mood: State Trait Anxiety Inventory (STAI) | Four nights, each night a week apart, spanning one month
  The STAI assesses anxiety and is composed of a state and a trait scale. Scores in either can range from 20 - 80, and higher scores indicate greater anxiety. Mean scores for healthy adult males of the state and trait scales are, respectively 35.7 (SD = 10.4) and 34.9 (SD = 9.2).
Awakening response: cortisol | Four mornings, each morning a week apart, spanning one month
  Salivary cortisol samples will be taken at regular intervals each morning in the lab to assess the awakening response. Higher values of cortisol concentrations indicate an stronger signal in this process of gaining alertness after sleep.
Awakening response: Psychomotor Vigilance Task (PVT) | Four mornings, each morning a week apart, spanning one month
  To assess behavioral response to awaking after sleep, a simple 10 minute reaction time task at the computer called the PVT will be administered. Typical reaction times for an adult are < 500 ms from stimulus presentation. Higher values will be expected for greater degree of sleep inertia after awakening.
Sleep inertia Questionnaire - Acute (SIQ - Acute) | Four mornings, each morning a week apart, spanning one month
  The SIQ - Acute assesses the subjective experience of the process of regaining alertness after waking from a sleep episode. Scores range from -66 to +66, higher scores indicating greater difficulty in regaining normal levels of alertness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Select An Option…, Switzerland